CLINICAL TRIAL: NCT06765382
Title: Association of Vitamin D Intake, and Associated Factors with Low Back Pain: a Retrospective Cohort Study
Status: Completed | Type: Observational
Sponsor: Mutah University (Other)
Responsible Party: Principal Investigator, Mohammad Abu-Jeyyab, Mutah University, Mutah University
Other Study IDs: 1502024; 1502024 (Other: Mutah University)
Record Dates: First submitted 2025-01-03; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2024-02

CONDITIONS: Vitamin D
Keywords: : Low back pain, Vitamin D, Pain, Disability, Oswestry low back disability questionnaire
MeSH Terms: conditions — Low Back Pain; Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
While there have been studies indicating a connection between insufficient levels of vitamin D and persistent low back pain (LBP), there is still a lack of definitive evidence. The primary objective of this study was to evaluate the correlation between vitamin D intake, and associated factors with chronic lower back pain.

ELIGIBILITY:
Inclusion Criteria:

* We included patients that were presented at our institute with chronic LBP and no associated comorbidities.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: We included patients that were presented at our institute with chronic LBP and no associated comorbidities.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Lower back pain | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Ibn Haytham Hospital, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No